CLINICAL TRIAL: NCT01424111
Title: Exploring Biomarkers for Depression
Status: Completed | Type: Observational
Sponsor: Wyss Institute at Harvard University (Other)
Collaborators: Massachusetts General Hospital (Other); Martinos Center for Biomedical Imaging (Other); Massachusetts Institute of Technology (Other)
Responsible Party: Sponsor
Other Study IDs: AMD-CS-0007
Record Dates: First submitted 2011-08-19; First posted 2011-08-26 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Major Depressive Disorder
Keywords: Biomarkers; Depression; Major Depressive Disorder; Escitalopram
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Escitalopram; Dexetimide

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Treatment: Those receiving an open-label, 10-20 mg/day, flexible-dose of escitalopram. The treatment period is 8 weeks long.
  Interventions: Drug: Escitalopram
- Healthy Control: Those not receiving treatment.
  Interventions: Other: Healthy Control

INTERVENTIONS:
Drug: Escitalopram — An open-label, 10-20 mg/day, flexible-dose of escitalopram will be administered to all subjects included in this study in the form of tablets. The treatment period is 8 weeks long.
  Other Names: Lexapro; Cipralex; Seroplex; Lexamil; Lexam
  Groups: Treatment
Other: Healthy Control — No Treatment
  Groups: Healthy Control

SUMMARY:
The purpose of this research is to explore objective biomarkers in voice, physiological, motor, and brain imaging signals that may one day be used to complement clinical evaluation and treatment of depression.

DETAILED DESCRIPTION:
The hypothesis for our work is that dynamical fluctuations of biological signals, such as, voice, video, pulse rate, oxygen saturation, skin temperature, skin conductivity, motor response, magnetoencephalography (MEG), and electroencephalography (EEG), are less complex during depressive than normal phases. There is a great need for objective biomarkers that may complement current clinical measures to help recognize depression, monitor its severity, and quantify the effect of interventions and recovery.

Data will be collected from 20 adult participants seeking outpatient treatment for depression at the Depression and Clinical Research Program at Massachusetts General Hospital (MGH), each participating for a total of approximately 9 weeks. For correlation of findings, data will also be collected from 20 subjects who take part in the healthy/control group. The healthy/control group will participate in a more limited study visit schedule over the course of 9 weeks, and will not be given any treatment. During study visits, the investigators will conduct recordings of voice, video, pulse rate, oxygen saturation, body temperature, skin conductivity, and motor movement at the Department of Psychiatry at MGH. In addition, each subject may participate in MEG, EEG, and Magnetic Resonance Imaging (MRI) brain imaging sessions at the Athinoula A. Martinos Center for Biomedical Engineering.

In order to collect relevant data and correlate findings with accepted clinical measures of depression severity and response to treatment, this study is conducted as a follow-up study in concert with a typical drug treatment protocol for Major Depressive Disorder (MDD). Specifically, our measurements will be made in conjunction with a standard of care drug treatment protocol using the antidepressant medication escitalopram, an FDA-approved selective serotonin re-uptake inhibitor (SSRI) commonly used to treat depression. The data will be collected over a period of approximately 9 weeks.

ELIGIBILITY:
Treatment Group Inclusion Criteria:

1. Men or women age 18-65;
2. Written informed consent;
3. Meet DSM-IV criteria (by Structured Clinical Interview for DSM-IV - SCID-I/P) for current major depressive episode (MDE);
4. Hamilton Rating Scale for Depression (HAM-D-17) baseline score ≥ 16.

Treatment Group Exclusion Criteria:

1. Subjects whose first language is not English;
2. In women, pregnancy, plans to conceive, or unwillingness to comply with birth control requirements;
3. Subjects with a baseline Clinical Global Impressions-Severity score of 6 or 7;
4. Subjects with suicidal ideation where outpatient treatment is determined unsafe by the clinician. These subjects will be immediately referred to appropriate clinical treatment;
5. Serious or unstable medical illness, including cardiovascular, hepatic, renal, respiratory, endocrine, neurologic or hematologic disease;
6. History of seizure disorder;
7. History or current diagnosis of the following DSM-IV psychiatric illness: organic mental disorder, schizophrenia, schizoaffective disorder, delusional disorder, psychotic disorders not otherwise specified, bipolar disorder, patients with mood congruent or mood incongruent psychotic features, patients with substance dependence disorders, including alcohol, active within the last 12 months;
8. Subjects with mood congruent or mood incongruent psychotic features;
9. Clinical or laboratory evidence of hypothyroidism;
10. Positive urine drug screen at evaluation visit;
11. Electro Convulsive Therapy (ECT) during the last year;
12. Subjects who have failed to respond during the course of their current major depressive episode to a trial of escitalopram (at least 40mg/day for six weeks or more)
13. History of intolerance to citalopram or escitalopram;
14. Subjects requiring excluded medications including antidepressants, anorexics, antiarrhythmics, and other psychotropic agents (including lithium, benzodiazepine sedatives, other sedatives, and anti-seizure medications), beta-blockers (such as metoprolol or propranolol) ketoconazole, itraconazole, fluconazole, erythromycin, omeprazole, cimetidine, dehydroepiandrosterone (DHEA), entacapone, hydroxytryptophan (5-HTP), ginkgo, St. John's Wort (hypercium), naratriptan, rizatriptan, sibutramine, zolmitriptan and warfarin (Coumadin).
15. Subjects who have failed two or more adequate antidepressant trials during the current Major Depressive Episode (MDE)

    If a subject is deemed eligible from the above criteria, there is additional exclusion criteria required to participate in Martinos Center study visits, listed below. Subjects meeting any of the below criteria will not be allowed to participate in visits to the Martinos Center.
16. Subjects of weight above 300 lbs. (limit for 1.5T Siemens Sonata whole body scanner used in MRI data acquisition);
17. History of significant head trauma (unconsciousness for 10 minutes or longer);
18. Surgical aneurysm clips;
19. Cardiac pacemaker;
20. Prosthetic heart valve;
21. Use of a neurostimulator;
22. Implanted pumps;
23. Cochlear implants;
24. Metal rods, plates, or screws in the body, or metal foil medical skin patches that cannot be removed;
25. IUD;
26. Previous head surgery;
27. Hearing aid;
28. Non-removable dentures, root canals, dental implants, bridges, and wires in the mouth;
29. Currently breastfeeding;
30. Meniere's Disease;
31. Metal (shiny) tattoos or metal body jewelry that cannot be removed;
32. Claustrophobia;
33. Abnormal hearing;
34. Glasses with vision correction greater than +/- 6 diopters.

Healthy/Control Group Inclusion Criteria:

1. Men or Women, ages 18-65;
2. Written informed consent;
3. QIDS-SR score of < 8 at Screening Visit;
4. Agrees to, and is eligible for, all biomarkers procedures (M/EEG, MRI, physiological recordings);

Healthy/Control Group Exclusion Criteria:

1. Subjects whose first language is not English;
2. Current or lifetime history for major depressive disorder, psychotic depression bipolar (I, II, or NOS) disorder, schizoaffective disorder, schizophrenia, or other Axis I psychotic disorder;
3. Meet DSM-IV criteria (by Structured Clinical Interview for DSM-IV - SCID-I/P) for current major depressive episode (MDE);
4. HAM-D-17 baseline score ≥ 8
5. Any current Axis I or Axis II diagnoses;
6. A woman who is pregnant or breastfeeding;
7. Meeting DSM-IV criteria for substance dependence in the last 6 months, except for nicotine, or substance abuse in the last 2 months;
8. Positive urine drug screen at evaluation visit;
9. Any current history for an unstable general medical condition (GMC) that requires hospitalization or deemed by investigator to be clinically significant;
10. Any current history for a moderate or severe acute or chronic medical condition that, based on the judgment of the PI or appropriate medical personnel would exclude the subject i.e. epilepsy, unstable hypothyroidism;

    If a subject is deemed eligible from the above criteria, there is additional exclusion criteria required to participate in Martinos Center study visits. Subjects meeting any of the below criteria will not be allowed to participate in visits to the Martinos Center:
11. Subjects of weight above 300 lbs. (limit for 1.5T Siemens Sonata whole body scanner used in MRI data acquisition);
12. History of significant head trauma (unconsciousness for 10 minutes or longer);
13. Surgical aneurysm clips;
14. Cardiac pacemaker;
15. Prosthetic heart valve;
16. Use of a neurostimulator;
17. Implanted pumps;
18. Cochlear implants;
19. Metal rods, plates, or screws in the body, or metal foil medical skin patches that cannot be removed;
20. IUD;
21. Previous head surgery;
22. Hearing aid;
23. Non-removable dentures, root canals, dental implants, bridges, and wires in the mouth;
24. Currently breastfeeding;
25. Meniere's Disease;
26. Metal (shiny) tattoos or metal body jewelry that cannot be removed;
27. Claustrophobia;
28. Abnormal hearing;
29. Glasses with vision correction greater than +/- 6 diopters.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients seeking treatment for Major Depressive Disorder at the Depression Clinical and Research Program at Massachusetts General Hospital. This study also enrolls a limited number of healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2011-08; Primary Completion 2017-10-14 (Actual); Study Completion 2017-10-14 (Actual)

PRIMARY OUTCOMES:
Objective Biomarkers | Participants will be followed for an expected average of 9 weeks of data collection.
  Objective biomarkers in voice, physiological, motor and brain imaging signals

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Nierenberg, MD, Principal Investigator — DCRP, Massachusetts General Hospital; Diana Young, Ph.D, Principal Investigator — Wyss Institute, Harvard University; Tommi Raij, MD, Ph.D, Principal Investigator — Martinos Center, Massachusetts General Hospital
Locations (1):
- Depression Clinical and Research Program, MGH, Boston, Massachusetts, United States